CLINICAL TRIAL: NCT02677714
Title: 99mTc-rhAnnexin V-128 Imaging of Apoptosis and Cardiotoxicity in Relationship to Ventricular Function in Patients With Early Stage Breast Cancer Receiving Doxorubicin-Based Chemotherapy
Brief Title: 99mTc-rhAnnexin V-128 Imaging and Cardiotoxicity in Patients With Early Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision based on strategic considerations
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAA-Annexin-05; CAAA113A42202 (Other: Novartis)
Record Dates: First submitted 2016-01-26; First posted 2016-02-09 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Doxorubicin Induced Cardiomyopathy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with breast cancer receiving chemotherapy (Experimental): After reconstitution and radiolabeling, 99mTc-rhAnnexin V-128 was administered as a single intravenous bolus of 350 MBq +/- 10% at baseline, after the 2nd cycle, after the 4th cycle and 12 weeks after AC chemotherapy.
  Interventions: Radiation: 99mTc-rhAnnexin V-128

INTERVENTIONS:
Radiation: 99mTc-rhAnnexin V-128 — Kit for the preparation of 99mTc-rhAnnexin V-128

SUMMARY:
This was a single center, proof-of-concept (PoC), Phase II study. Patients with histologically confirmed early stage (Stage I, II or III) HER-2 negative breast cancer and scheduled to receive doxorubicin-based (neo)adjuvant therapy to be followed by paclitaxel or docetaxel as per clinical practice. The planned doxorubicin-based chemotherapy treatment consisted of doxorubicin 60 mg/m2 in combination with cyclophosphamide 600 mg/m2 (AC) intravenous (IV) every 2 or 3 weeks for 4 cycles. Patients were scheduled for CMRI and 99mTc-rhAnnexin V-128 imaging (planar and SPECT / CT) at the following visits:

1. Screening/baseline, i.e. 2 weeks prior to initiating AC treatment (Visit 1)
2. After the 2nd and before the 3rd cycle of AC treatment (Visit 2)
3. After the 4th cycle of AC treatment and within 2 weeks (Visit 3)
4. At 12 weeks after the 4th cycle of AC treatment (Visit 4). The imaging procedures were conducted and analyzed. Bloodwork for cardiotoxicity biomarkers (troponin, N terminal pro B-type natriuretic peptide [NT-proBNP]) was performed at each visit.

DETAILED DESCRIPTION:
Overall, it was planned to recruit 30 adults with early stage breast cancer. The first 10 patients were to be enrolled in the PoC phase of the study to assess the potential of 99mTc-rhAnnexin V-128 in terms of imaging quality, uptake and medical relevance. Based on the results of the first 10 patients, the DMC was to decide whether to terminate the study or continue to the Phase II and enroll the next 20 planned patients. The maximum study duration was 26 (±4) weeks per patient (including the screening and follow-up periods).

The sponsor decided to terminate the study earlier than planned due to strategic decisions to focus the AAA development portfolio on oncology theragnostics and not based on safety concerns.

ELIGIBILITY:
Inclusion criteria:

1. Females >= 18 years of age with histologically confirmed early stage (Stage I, II or III) HER-2 negative breast cancer and planned for (neo)adjuvant doxorubicin-based chemotherapy (AC every 2 or 3 weeks x 4 cycles)
2. Eastern Cooperative Oncology Group Status (ECOG) ≤ 2
3. Able and willing to comply with the study procedures

Exclusion criteria:

1. Pregnancy or lactation
2. Moderate or severe valvular stenosis or regurgitation
3. History of atrial fibrillation or flutter
4. History of any disease or relevant physical or psychiatric condition which may interfere with the study objectives at the investigator judgment
5. Know hypersensitivity to the investigational product (IP) or any of its components
6. Prosthetic valve or pacemaker
7. Claustrophobia or inability to lie still in a supine position
8. Contraindication(s) to the CMRI procedure
9. Participation in another clinical trial within 4 weeks before study inclusion, except for patients who have participated or who are currently participating in a study without any study drug administration
10. Unwillingness to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in Canada.
Groups:
- 99mTc-rhAnnexin V-128 (Part I / Proof of Concept); 99mTc-rhAnnexin V-128 (Part II / Phase II): After reconstitution and radiolabeling, 99mTc-rhAnnexin V-128 was administered as a single intravenous bolus of 350 MBq +/- 10% at baseline, after the 2nd cycle, after the 4th cycle and 12 weeks after AC chemotherapy.
Period: Overall Study
Arm/Group | 99mTc-rhAnnexin V-128 (Part I / Proof of Concept) | 99mTc-rhAnnexin V-128 (Part II / Phase II)
Started (All enrolled patients who were dosed were included in both the full analysis set (FAS) and the safety set) | 12 | 2
Completed | 10 | 2
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 99mTc-rhAnnexin V-128 (Part I / Proof of Concept) | 99mTc-rhAnnexin V-128 (Part II / Phase II) | Total
Number analyzed (Participants) | 12 | 2 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (9.3) | 39.0 (0.0) | 52.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 14
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 1 | 0 | 1
  Caucasian | 11 | 0 | 11
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part I / Proof of Concept (PoC): Number of Participants Evaluated for Imaging Feasibility
Description: The feasibility of imaging apoptotic activity using 99mTc-rhAnnexin V-128 was assessed in the first 10 patients who enrolled and completed the PoC phase of the study by the data monitoring committee (visual image review and consensus). The three reviewers of the DMC did an independent visual assessment of the images using a 1 to 4 point grading system: each observer reviewed the images of each patient and scored either 1 or 2 (uptake was less than or equal to blood pool), these images were considered normal; 3 was equivocal and four equalled abnormal. Only descriptive analysis performed.
Time Frame: Day 0 (Baseline)
Population: Full Analysis Set population (FAS). Only the first 10 participants who enrolled and completed the PoC phase of the study were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 99mTc-rhAnnexin V-128 (Part I / Proof of Concept)
Number analyzed (Participants) | 10
Participants | 10

2. Secondary Outcome: 99mTc-rhAnnexin V-128 Myocardial Uptake
Description: Single-Photon Emission Computed Tomography (SPECT)/Computed Tomography (CT) scans of the thorax were acquired with a dual head SPECT/CT gamma camera with low-energy high-resolution collimators at 1 and 2 hours post-injection at each collection time point and were to be compared to Baseline. Myocardial uptake was measured from regions of interest (ROIs) placed over the myocardium on the SPECT images coregistered with the corresponding CT images for anatomic delineation. Myocardial uptake was expressed either in absolute units (% injected dose/g) or as a standardized uptake value (SUV). Only descriptive analysis performed.
Time Frame: 60 and 120 minutes post injection at: Day 0 (Baseline), Visit 2 (After the 2nd and before the 3rd cycle of doxorubicin), Visit 3 (After the 4th cycle of doxorubicin and within 2 weeks), Visit 4 (12 weeks after the 4th cycle of doxorubicin)
Population: Full Analysis Set population (FAS). Only the participants who completed the 4 chemotherapy treatment cycles and underwent all study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of injected dose/g
Arm/Group | 99mTc-rhAnnexin V-128 (Part I / Proof of Concept) | 99mTc-rhAnnexin V-128 (Part II / Phase II)
Number analyzed (Participants) | 10 | 2
percentage of injected dose/g
  Day 0 - 60 mins after injection | 0.0035617 (0.0051846) | 0.0003306 (0.0004675)
  Day 0 - 120 mins after injection | 0.0024177 (0.0036831) | 0.0002125 (0.0003004)
  Visit 2 - 60 mins after injection | 0.0043825 (0.0067130) | 0.0008123 (0.0011487)
  Visit 2 - 120 mins after injection | 0.0029255 (0.0045063) | 0.0004827 (0.0006826)
  Visit 3 - 60 mins after injection | 0.0018097 (0.0011105) | 0.0000512 (0.0000723)
  Visit 3 - 120 mins after injection | 0.0016232 (0.0008994) | 0.0002995 (0.0004236)
  Visit 4 - 60 mins after injection | 0.0020756 (0.0008986) | 0.0010116 (0.0014306)
  Visit 4 - 120 mins after injection | 0.0018475 (0.0005084) | 0.0006692 (0.0009463)

3. Secondary Outcome: Changes in Left Ventricular (LV) Function
Description: The worsening of LV function was to be assessed by comparing cardiac magnetic resonance imaging (CMRI) left ventricular ejection fraction (LVEF) after the 2nd and the 4th cycle of doxorubicin/cyclophosphamide chemotherapy (AC) treatment and after 12 weeks of the last dose of doxorubicin compared to Baseline. Only descriptive analysis performed.
Time Frame: Day 0 (Baseline), Visit 2 (After the 2nd and before the 3rd cycle of doxorubicin), Visit 3 (After the 4th cycle of doxorubicin and within 2 weeks), Visit 4 (12 weeks after the 4th cycle of doxorubicin)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | 99mTc-rhAnnexin V-128 (Part I / Proof of Concept) | 99mTc-rhAnnexin V-128 (Part II / Phase II)
Number analyzed (Participants) | 10 | 2
Percent
  Day 0 | 66.8 (5.37) | 64.0 (2.83)
  Visit 2 | 66.3 (6.07) | 60.5 (0.71)
  Visit 3 | 64.0 (4.57) | 65.0 (1.41)
  Visit 4 | 63.6 (4.22) | 62.5 (2.12)

4. Secondary Outcome: Changes in the Cardiotoxicity Biomarkers (Troponin and NT-proBNP)
Description: The differences of LV function after the 2nd and the 4th cycle of doxorubicin/cyclophosphamide chemotherapy (AC) treatment and after 12 weeks of the last dose of doxorubicin compared to Baseline were to be correlated with the changes in cardiotoxicity biomarkers: Troponin and N Terminal pro B-type Natriuretic Peptide (NT-proBNP). Only descriptive analysis performed.
Time Frame: as for outcome 3
Population: Full Analysis Set population (FAS). For each parameter, only participants with a value at both baseline and post baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | 99mTc-rhAnnexin V-128 (Part I / Proof of Concept) | 99mTc-rhAnnexin V-128 (Part II / Phase II)
Number analyzed (Participants) | 12 | 2
ng/L
  Troponin - Day 0 | 0.015 (0.001) | 0.015 (0.000)
  Troponin - Visit 2: number analyzed (Participants) | 9 | 2
  Troponin - Visit 2 | 0.019 (0.010) | 0.015 (0.000)
  Troponin - Visit 3: number analyzed (Participants) | 10 | 2
  Troponin - Visit 3 | 0.025 (0.019) | 0.015 (0.000)
  Troponin - Visit 4: number analyzed (Participants) | 10 | 2
  Troponin - Visit 4 | 0.060 (0.088) | 0.028 (0.018)
  NT-proBNP - Day 0 | 49.6 (27.50) | 60.0 (63.64)
  NT-proBNP - Visit 2: number analyzed (Participants) | 10 | 2
  NT-proBNP - Visit 2 | 271.8 (399.76) | 104.0 (86.27)
  NT-proBNP - Visit 3: number analyzed (Participants) | 10 | 2
  NT-proBNP - Visit 3 | 123.7 (66.30) | 85.0 (49.50)
  NT-proBNP - Visit 4: number analyzed (Participants) | 10 | 2
  NT-proBNP - Visit 4 | 123.6 (89.27) | 74.0 (29.70)

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent until the last study-related procedure (up to 12 weeks)
Arm/Group | 99mTc-rhAnnexin V-128 (Part I / Proof of Concept) | 99mTc-rhAnnexin V-128 (Part II / Phase II)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/2
Other Adverse Events (participants affected / at risk) | 10/12 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 99mTc-rhAnnexin V-128 (Part I / Proof of Concept) (N=12) | 99mTc-rhAnnexin V-128 (Part II / Phase II) (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (Gastrointestinal disorders) | 0 | 1
Carbuncle (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 99mTc-rhAnnexin V-128 (Part I / Proof of Concept) (N=12) | 99mTc-rhAnnexin V-128 (Part II / Phase II) (N=2)
Palpitations (Cardiac disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 1 | 0
Dysgeusia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 7 | 2
Febrile neutropenia (General disorders) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Insomnia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Sleep disorder due to general medical condition, insomnia type (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Skin candida (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the early termination of the trial and the fact that only 2 patients were enrolled in the Phase II of the study, the efficacy endpoints of the trial were not addressed (summary statistics were not performed).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-03-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT02677714/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT02677714/SAP_001.pdf